CLINICAL TRIAL: NCT02653469
Title: Pulse Pressure Variation With Augmented Ventilation to Predict Fluid Responsiveness in the Patients Undergoing Open Laparotomy Surgery
Brief Title: Augmented Pulse Pressure Variation to Predict Fluid Responsiveness in Open Laparotomy
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Assistant professor, Samsung Medical Center
Other Study IDs: SMC 2015-06-015
Record Dates: First submitted 2015-10-20; First posted 2016-01-12 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Gynecologic Neoplasms; Abdominal Neoplasms
MeSH Terms: conditions — Genital Neoplasms, Female; Abdominal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Augmented ventilation with fluid loading: This is an observational study and as a diagnostic intervention, subjects in the study would receive mechanical ventilation with augmented tidal volume of 12ml/kg for 2min. Augmented ventilation is performed when the patient's PPV is within grey zone (9-13%). The investigators perform this procedure to every patients and do not assigh this intervention to the subjects of the study. Then, 6ml/kg of ballanced crystalloid loading will be infused to every patient.
  Interventions: Other: Augmented ventilation; Other: Fluid loading

INTERVENTIONS:
Other: Augmented ventilation — When the patient's PPV is within grey zone, patient's tidal volume is maintained with augmented tidal volume of 12 ml/kg (from normal ventilation of 8ml/kg) for 2min duration.
Other: Fluid loading — We record the stroke volume index (SVI) values before and after volume expansion with 6ml/kg of balanced crystalloid
  Other Names: Balanced crystalloid infusion

SUMMARY:
Pulse pressure variation (PPV) is a well-known and widely used dynamic preload indicator based on heart-lung interaction to predict fluid responsiveness. Generally, patients are considered to be fluid-responsive when the PPV value larger than 11-13%. However, several previous researches demonstrated that there is a zone of uncertainty (grey zone) in PPV. To predict fluid-responsiveness accurately in the patients with PPV within grey zone (9-13%), the investigators would evaluate the augmented PPV using augmented ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective open laparotomy surgery.

Exclusion Criteria:

* Irregular heart beats,
* cardiac arrhythmia,
* moderate or severe valvular heart disease,
* preoperative left ventriular ejection fraction less than 40%,
* moderate t severe obstructive pulmonary disease,
* preoperative need of inotropics infusion,
* preoperative serum Cr > 1.3ml/dl,
* moderate to severe renal or liver disease,
* acute lung injury or acute lung problem,
* coexisting open chest condition,
* severe bradycardia,
* patients with spontaneous breathing

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective open laparotomy surgery.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Augmented PPV (Pulse Pressure Variation) to predict fluid responsiveness | within 2 min from augmented ventilation
  Augmented ventilation (12ml/kg) will be performed when the participant's PPV is within grey zone (9-13%). PPV value will be collected automatically by Intelivue philips patient monitor. Percentage changes in stroke volume index by EV1000 according to fluid loading were used as principal indicators of fluid responsiveness. Patients were classified as responders or non-responders when increases in SVI were ≥ 10% or <10% after volume loading (crystalloid iv 6ml/kg). To test the abilities of augmented PPV to predict fluid responsiveness, areas under the receiver operating characteristics (ROC) curves of the responders [area under the curve (AUC) = 0.5: no better than chance, no prediction possible; AUC = 1.0: best possible prediction] will be calculated.

SECONDARY OUTCOMES:
Conventional baseline PPV to predict fluid responsiveness | when patients PPV in grey zone, before augmented ventilation
  PPV value will be collected automatically by Intelivue philips patient monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Min JJ, Gil NS, Lee JH, Ryu DK, Kim CS, Lee SM. Predictor of fluid responsiveness in the 'grey zone': augmented pulse pressure variation through a temporary increase in tidal volume. Br J Anaesth. 2017 Jul 1;119(1):50-56. doi: 10.1093/bja/aex074. PMID 28974059